CLINICAL TRIAL: NCT05988749
Title: American Heart Association Digital Home Remote Monitoring for Heart Failure
Brief Title: Digital Remote Home Monitoring for Heart Failure
Acronym: ADHERE-HF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Nicholas Hendren, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2023-0529
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure, Systolic
Keywords: remote home monitoring; heart failure; guideline directed medical therapy
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:2 fashion to usual care versus usual care plus the American Heart Association's Digital Solution by dice roll.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device (Experimental): Participants will receive usual care or usual care plus the American Heart Association's Digital Solution in patients with HFrEF. The Solution is a combination of the AHA/CHTI HF CarePlans and Education Content, delivered through and combined with the Biofourmis Platform.
  Interventions: Other: Biofourmis Digital Platform
- Routine Care (No Intervention): Routine care for heart failure management

INTERVENTIONS:
Other: Biofourmis Digital Platform — The intervention is a combination of the American Heart Association's Digital Heart Failure CarePlans and Education Content, delivered through and combined with the Biofourmis Platform. Patients enrolled in this arm will wear the device for 90 days and provide data to the participant's care team.
  Other Names: American Heart Association's Digital Heart Failure CarePlans and Education Content
  Arms: Device

SUMMARY:
We will enroll 150 adult participants with systolic heart failure into the ADHERE-HF trial. The study will randomize participants in a 1:2 fashion to usual care or usual care plus the American Heart Association's Digital Solution for 90 days. This wearable device and careplan package is hypothesized to improve rates of guideline directed heart failure medical care for participants.

DETAILED DESCRIPTION:
Background/Rationale:

Guideline-directed medical therapy (GDMT) is a cornerstone of the management of individuals with heart failure with reduced ejection fraction (HFrEF). Patients on optimal heart failure pharmacotherapy experience higher survival rates and fewer heart failure hospitalizations compared with subjects not on these medications [1,2]. Furthermore, optimal compliance with these treatments among patients with heart failure is associated with fewer have fewer emergency department visits, fewer hospital admissions, shorter lengths of hospital stay, and lower risk of death [3,4].

Despite very strong evidence for these treatments, a substantial proportion of eligible subjects with HFrEF are not on GDMT at optimal dosages. Data from the CHAMP-HF registry demonstrate that fewer than one in four HFrEF subjects are on all three of GDMT medications - beta-blockers; angiotensin-converting enzyme inhibitor (ACEi)/angiotensin II receptor blocker (ARB), or angiotensin receptor neprilysin inhibitor (ARNI); and mineralocorticoid receptor antagonist (MRA) - and only 1% were receiving target doses of all three medications [4]. Published data for both UT-Southwestern and Parkland Health System have demonstrated that rates of GDMT are above national averages but remain suboptimal with significant room for improvement.

Successful interventions to increase the number of subjects of prescribed GDMT at optimal doses often have included multidisciplinary heart failure clinics that include advanced practice providers and/or pharmacists with frequent visits [5,6]. However, such strategies are resource-intensive and are not widely applicable to heart failure management outside of specialized heart failure clinics. Health systems, such as Parkland Health System and UT-Southwestern, have also considered and purchased remote home monitoring programs for patients with systolic heart failure to try to improve prescription rates of GDMT. However, few studies have evaluated the impact of remote home monitoring on rates of GDMT in highly diverse patient populations or patients with increased socioeconomic risk.

As such, there is a crucial unmet need to implement highly effective GDMT titration strategies in heart failure populations with increased socioeconomic risk and the effects of remote monitoring systems to improve GDMT are not well known.

To address this gap in knowledge, we will leverage the large, multiethnic heart failure populations followed in two health systems, UT-Southwestern and Parkland Health System. Using these racially and ethnically diverse patient populations, we will test our central hypothesis that the AHA Digital Platform will improve outcomes in patients with HFrEF by managing the initiation and titration of heart failure GDMT in comparison with clinical care. The purpose of this study is to assess the effectiveness of the remote monitoring AHA Digital Platform to improve initiation and titration of GDMT in addition to traditional clinical encounters. The effective comparison will be to the current standard of care for heart failure used in the respective clinical sites.

The AHA Digital platform integrates data from remote wireless vital signs collection devices and an investigational wearable health device to recommend optimal titration of GDMT in subjects with heart failure with reduced ejection fraction (HFrEF) subjects or HFrEF subjects on suboptimal doses of GDMT. The platform uses a proprietary algorithm to interpret the remote vitals data collected and presents titration recommendations back to the healthcare provider (HCP) via a HCP mobile App for subjects randomized to the Intervention Arm at his/her site. Vitals data and relevant HF educational materials are simultaneously presented to the subject via a Patient App. Data from an investigational wearable health device is also provided to both the HCP and subject, however no care decisions are made with the data from this device. The HCP is also alerted to changes in status of the respective participating trial subjects via the HCP App and can see aggregated information and further visualize the status of all subjects enrolled in his/her center via an online web portal.

Hypothesis We hypothesize that use of the AHA Digital Solution in a real-world, multi-site, randomized, outpatient study will improve rates and does of optimal Guideline-Directed Medical Therapy (GDMT) for patients with heart failure with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-year-old adults with a clinical diagnosis of heart failure AND a left ventricular ejection fraction ≤40% by transthoracic echocardiogram or cardiac MRI within 12 months prior to enrollment.

Exclusion Criteria:

* Patients who are pregnant.
* Patients who do not have a smartphone or access to the Internet
* Prisoners or refugees.
* Patients who are homeless or have unstable housing.
* Unable or unwilling to consent or use study related materials.
* On-going cocaine, methamphetamine, opioid, alcohol, or other illicit substance abuse as determined by the study PI.
* Not fluent in English or Spanish.
* Students or trainees at UT-Southwestern or Parkland Health System.
* Enrolled or considering hospice.
* Recent or home inotropic therapy, or heart transplant evaluation.
* Survival anticipated <6 months.
* End-stage renal disease, receiving dialysis or eGFR ≤30 mL/min/1.73m2
* Non-Texas resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
GDMT score | 0-90 days
  Change in GDMT score from between the intervention and control arm.

SECONDARY OUTCOMES:
Hospitalized days | 0-90 days; 0-180 days
  Number of days hospitalized between the intervention and control arm
Emergency room visits | 0-90 days; 0-180 days
  Number of emergency room visits between the intervention and control arm
GDMT score | 0-180 days
  Change in GDMT score from between the intervention and control arm.
Change in KCCQ-12 score | day 0-90 and 0-180
  Change in overall and subdomain KCCQ-12 scores from between the intervention and control arm
Visual analog score change | day 0-90
  Change in visual analog scores from between the intervention and control arm
Optimal GDMT dosing | 0-90 days, 0-180 days
  Difference between the intervention and control arm in the percentage of subjects on optimal doses of GDMT

OTHER OUTCOMES:
Patient encounters | 0-90; 0-180 days
  Number of clinical patient encounters (phone, Mychart, clinic visit)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hendren, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health & Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No